CLINICAL TRIAL: NCT02443090
Title: An 8-Week Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Oral Fispemifene for the Treatment of Sexual Dysfunction in Hypogonadal Men
Brief Title: Safety and Efficacy Study of Oral Fispemifene for the Treatment of Sexual Dysfunction in Hypogonadal Men
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NexMed (U.S.A.), Inc. (subsidiary of Apricus Biosciences, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NM-F15-202
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Secondary Hypogonadism; Sexual Dysfunction; Erectile Dysfunction
Keywords: secondary hypogonadism; sexual dysfunction; erectile dysfunction
MeSH Terms: conditions — Hypogonadism; Sexual Dysfunction, Physiological; Erectile Dysfunction | interventions — fispemifene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fispemifene 450 mg (Experimental): Fispemifene capsules will be taken orally each morning immediately after eating a meal
  Interventions: Drug: fispemifene
- Placebo (Placebo Comparator): Placebo capsules will be taken orally each morning immediately after eating a meal
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: fispemifene
  Arms: Fispemifene 450 mg
Other: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of fispemifene in men with secondary hypogonadism and sexual side effects.

DETAILED DESCRIPTION:
This phase 2 study is a double-blind, placebo controlled, parallel arm study with a 4 week run-in and an 8-week treatment period. It will assess the safety and tolerability of fispemifene, and the effects of treatment on the sexual side effects seen in this patient population using PRO endpoints.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of secondary hypogonadism
* Mild to moderate erectile dysfunction
* Ability to read, understand and complete diaries and questionnaires
* Ability to safely make sexual attempts during the course of the study

Exclusion Criteria:

* Primary hypogonadism
* Hypogonadism as a result of surgery, trauma, tumors or radiation of the hypothalamus or pituitary
* History or current diagnosis of breast cancer, prostate cancer and/or PSA level above ≥3.5 ng/mL
* Poorly controlled blood pressure, type 2 diabetes, thyroid disease; sleep apnea
* Elevated prolactin level
* Hemoglobin >17 g/dL or Hematocrit >50%
* Use of transdermal or oral testosterone within 4 weeks, intramuscular testosterone therapy within 6 weeks, and testosterone pellets within 6 months prior to Screening and at any time throughout the study
* Use of another SERM or past participation in a trial with Fispemifene
* Use of medications known to alter the HPG axis
* Clinically significant findings on physical exam, screening labs, or other findings which would prevent safe participation in the study
* Participation in another clinical study in the last 30 days

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in IIEF-EF (International Index of Erectile Function - erectile function domain) score | 8 weeks
  Change in the IIEF-EF (International Index of Erectile Function - erectile function domain) score from Randomization to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Troupin, MD, MBA, Study Director — NexMed (U.S.A.), Inc.
Locations (16):
- United States (16):
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - San Diego Clinical Trials, San Diego, California
  - Genesis Research LLC, San Diego, California
  - Meridien Research, Bradenton, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - Premier Urology Associates, LLC, dba AdvanceMed Research, Lawrence, New Jersey
  - The Urological Institute of Northeastern New York, Albany, New York
  - AccuMed Research Associates, Garden City, New York
  - Bruce R. GIlbert, MD, PhD, PC, Great Neck, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Volunteer Research, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Physicians' Research Options LLC, Draper, Utah
  - Clinical Research Associates of Tidewater, Inc., Norfolk, Virginia